CLINICAL TRIAL: NCT03997773
Title: Face-it: A Health Promotion Intervention for Women With Prior Gestational Diabetes and Their Families - A Randomised Controlled Trial
Brief Title: Face-it: Health Promotion for Women With Prior Gestational Diabetes
Acronym: Face-it
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Steno Diabetes Center Odense (Other); Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Aarhus Municipality, Denmark (Other); Odense Municipality (Unknown); Copenhagen Municipality, Denmark (Other Government); Liva Healthcare A/S (Unknown)
Responsible Party: Principal Investigator, Helle terkildsen Maindal, Professor, Senior Researcher, MPH, PhD, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: StenoDC
Record Dates: First submitted 2019-05-29; First posted 2019-06-25 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Gestational Diabetes; Type 2 Diabetes Mellitus; Quality of Life
Keywords: Gestational Diabetes; Type 2 Diabetes; Family Intervention; Denmark; Health Promotion; Postpartum Intervention; Quality of Life; Wellbeing
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Two-arm parallel design RCT with women with prior GDM as the unit of randomisation comparing a health promotion intervention with a usual care group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Will receive the intervention
  Interventions: Behavioral: Face-it Intervention
- Usual care (No Intervention): Will receive usual care - will be the control group

INTERVENTIONS:
Behavioral: Face-it Intervention — The Face-it intervention is a health promotion intervention consisting of 3 major components: 1) active involvement of health visitors, 2) digital health technology and coaching, and 3) a structured cross-sectoral communication system in the healthcare system. The intervention will begin at time approx. 3 months (after the baseline data collection, i.e. 10-14 weeks postpartum), and continues until 12 months
  Arms: Intervention

SUMMARY:
This project focuses on evaluating a health promotion intervention among families where the mother has prior gestational diabetes mellitus (GDM) in the first year after delivery. The intervention focuses on the individual, family and health system levels. The aim is to increase quality of life and reduce the risk of type 2 diabetes among women with prior GDM and their families.

DETAILED DESCRIPTION:
Face-it: A Health Promotion Intervention for Women with Prior Gestational Diabetes and their Families

AIM: The aim of the Face-it project is to increase quality of life and reduce the risk of type 2 diabetes (T2DM) among women with prior gestational diabetes mellitus (pGDM) and their families.

BACKGROUND: Women with pGDM are at high risk of developing type 2 diabetes. Partners and offspring of women with GDM are also at elevated risk of developing type 2 diabetes and related cardiometabolic conditions. Thus, not only are women with prior GDM at high risk of T2DM and related cardiometabolic conditions, their children and spouses are as well. Since the cumulative incidence of T2DM increases substantially within the first five years after delivery (Kim et al. 2002) there is a strong interest in identifying feasible and effective interventions in this time-period. Evidence from the state-of-the-art Diabetes Prevention Program suggests that intensive lifestyle intervention can reduce the risk of T2DM among women with pGDM (Ratner et al. 2008). However, sustainable changes in such behaviours are difficult and many women do not follow lifestyle recommendations after delivery (Stage et al. 2004). Given the highly elevated risk in this group, this is a substantial missed opportunity for health promotion aimed at prevention of T2DM for not only the mother, but the entire family. It is vital that efforts are based on a thorough understanding of the barriers to health promoting behaviours and involve carefully tailored solutions to overcome these barriers. The investigators hypothesise that a health promotion intervention that focuses on enhancing motivation, health literacy, action competences and social involvement in women with pGDM and their families will reduce diabetes risk and improve quality of life.

DESIGN: Face-it is a two-arm parallel-group randomised clinical trial with women as the unit of randomization comparing a health promotion intervention with a usual care control group.

PARTICIPANTS, RECRUITMENT AND ELIGIBILIGY: Women with pGDM will be recruited from obstetric departments at Aarhus University Hospital (AUH), Odense University Hospital (OUH) or Rigshospitalet (RH) around 24-40 weeks of pregnancy by a health care professional. To be eligible for enrolment into the study, women should also be able to provide written informed consent in Danish. Exclusion criteria is that the participants may not be participating in other postpartum intervention trials with a possible impact on the Face-it trial. Women with diabetes identified at baseline will be excluded. Partners of women and the new-born offspring are also invited to participate in the study. Informed consents are obtained from 1) woman and new-born offspring, including permission to obtain information from the medical record and blood samples for research biobank (woman only), 2) from partner, including blood samples for research biobank. A separate consent 3) is obtained for collection of blood for future biobank. In case of non-participation in the study, women are asked for consent to collect information from the medical record including health characteristics of woman and offspring related to pregnancy and birth.

SAMPLE SIZE AND RANDOMISATION: Based on prior studies, a mean difference in BMI after 1 year between the intervention and control groups for the women of -1.0 kg/m2 and standard deviation of 2.5 is expected. A sample size of 225 women will be required to detect such a difference in BMI when using a 2:1 randomisation procedure, a power of at least 80% and type 1 error of 5% (two-sided). The sample size increases to 460 women to allow for assuming 30% loss to follow-up between baseline and follow-up and another 30% will withdraw during the prolonged period from recruitment to baseline data collection and randomisation.

1/3 of participants will be randomised to the control group and 2/3 to the intervention group. The randomization procedure has been generated by an independent statistician and will be in blocks of 6/9/12/15 with a separate randomization at each of the three recruitment locations. Allocation will be concealed from both the participant and the investigators, who have the clinical and research responsibility, until baseline data have been collected, eligibility confirmed, and participation accepted. However, neither participants nor the investigators will be blinded to the participants intervention or control status after this point, but the status will be blinded for the analyst. A randomization list will be kept securely at the study site by an investigator with clinical responsibility. Both the intervention and usual care group will be part of the evaluation of the Face-it trial and therefore invited to baseline and follow-up clinical examinations. Participants will be informed by a research assistant about whether they have been allocated to the control or intervention group.

INTERVENTION: The intervention has been developed in a thorough and iterative co-creation process with health care providers and families, where the mothers has pGDM to ensure that it is carefully tailored to the needs and challenges of the target group and enhance its sustainability. The three major components of the intervention are: 1) Health visitors as the core healthcare providers, 2) digital health technology, and 3) a structured cross-sectoral communication system in the healthcare system.

CONTROL: Participants in the control group will receive usual care practice, including recommended glucose control measures 3 months and one year after birth. Participants will receive advice about a healthy lifestyle according to the national recommendations from the Danish Health and Medicines Authority . Participants in the control group will be invited to participate in the health examination at baseline and follow-up and thereby obtain information about own health when attending the two clinical examinations.

STUDY PROCEDURES AND DATA COLLECTION: There are two study visits planned for each participant (women with pGDM, her partner and baby). Visit 1 (baseline) will take place 10-14 weeks postpartum. Visit 2 (follow-up) will take place around 12 months after delivery. The measurements taken at the visits are dependent on whether the participant is a women with pGDM, partner or offspring.

* 75g oral glucose tolerance test (OGTT) with measurements of glucose and insulin at 0, 30 and 120 minutes (women with pGDM only)
* Blood samples including fasting glucose, insulin secretion and insulin sensitivity Index, hbA1c, plasma lipids/ triglycerides, total cholesterol, HDL, LDL (women with pGDM and partners)
* Physical measures. Investigations on women with pGDM and their partners will include BMI, height, weight, waist- and hip circumference, body fat, blood pressure.
* Physical measures on offspring will include height, weight, abdominal- and head circumference (at one-year follow-up).
* Questionnaire. Detailed information will be collected about socio-demographic and -economic details, dietary-, physical activity-, and sleep patterns; quality of life, stress, depression, self-perceived health, health literacy, motivation for behaviour change, social support, self-efficacy, risk perception and knowledge about diabetes risk in women with pGDM and their partners. Information about obstetric history and breastfeeding will also be collected from women with pGDM
* Objective measures of physical activity and sedentary patterns (subgroup)

ELIGIBILITY:
Inclusion Criteria:

* Women with a GDM diagnosis according to current Danish guidelines (2h oral glucose tolerance test ≥9.0mmol/l)
* Women with a GDM diagnosis should also be attending and giving birth at the obstetric departments at either Aarhus University hospital, Odense University Hospital or Rigshospitalet
* Partner or infant of women with a GDM diagnosis
* Able to provide written informed consent in Danish

Exclusion Criteria:

* Concomitant participation in other postpartum intervention trial with a possible impact on the participation in the face it trial

Withdrawal Criteria:

* Participant's withdrawal of the informed consent
* Safety concerns, judged by the investigator
* Non-compliance with the protocol, judged by the investigator
* Woman with pGDM being diagnosed with type 1 or type 2 diabetes before or during the first examination (baseline data collection visit)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Measured at baseline and at follow-up 1 year after delivery
  To assess changes in BMI, height and body weight will be measured, and calculated kg/m2
Change in quality of life | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire. Quality of life will be measured using the 12-item Short Form Health Survey (SF-12v2). Summary score will be calculated for the mental health domain. The SF-12 summary score ranges from 0 to 100, with higher scores representing better self-reported quality of life/health.

SECONDARY OUTCOMES:
Change in fasting glucose | Measured at baseline and at follow-up 1 year after delivery
  Fasting glucose (mmol/L)
Change in HDL and triglycerides | Measured at baseline and at follow-up 1 year after delivery
  Blood samples will be drawn after an overnight fast and will include measures of lipids
Change in well-being | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire. Well-being will be measured with The WHO-Five Well-being Index (WHO-5). An individual score between 0 (worst possible ) and 100 (best possible) is calculated based on the replies to the five questions in the questionnaire.
Change in self-perceived health | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire. Self-perceived Health will be measured using the question "in general, would you say that your health is excellent, very good, good, fair, or poor?".
Change in stress | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire. Stress will be measured with the Perceived Stress Scale (PSS). Individual scores on the PSS ranges from 0 (lowest possible perceived stress level) to 40 (highest possible perceived stress level).
Change in anxiety | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire. Anxiety will be measured with the General Anxiety Disorder (GAD-7) scale. Individual scores on the GAD-7 ranges from 0 (lowest possible anxiety level) to 21 (highest possible anxiety level).
Change in dietary patterns | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire. Dietary patterns will be measured using the Dietary Quality Score (DQS-2017). The score is based on questions regarding intake of fruit, vegetables, fish and fats and is rated on a scale from 0 to 8, with 8 being the most optimal diet.
Change in moderate to vigorous physical activity patterns | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire. Physical activity will be measured using adapted version of the International Physical Activity Questionnaire (IPAQ) short form. Physical activity levels will be measured in minutes per week.

OTHER OUTCOMES:
Change in waist- and hip circumference in women with prior GDM | Measured at baseline and at follow-up 1 year after delivery
  Waist circumference will be measured halfway between the lowest point of the costal margin and highest point of the iliac crest; whereas hip circumference will be measured at the level of the greater femoral trochanter. Both will be measured to the nearest 0.5 cm.
Change in body fat% in women with prior GDM | Measured at baseline and at follow-up 1 year after delivery
  Body fat% will be measured using body impedance
Differences in %weight change | At follow-up 1 year after delivery
  Weight will be measured at baseline and 1 year after delivery, and the %weight change calculated
Change in 2h glucose | Measured at baseline and at follow-up 1 year after delivery
  After 2h OGTT
Change in HbA1c (mmol/mol) | Measured at baseline and at follow-up 1 year after delivery
  HbA1c measured in fasting blood sample
Change in fasting and 2h insulin (pmol/L) | Measured at baseline and at follow-up 1 year after delivery
  Measure in fasting blood sample and after 2h OGTT
Changes in HOMA-IR and HOMA-b | Measured at baseline and at follow-up 1 year after delivery
  Will be calculated based on the glucose and insulin measurements
Change in blood pressure | Measured at baseline and at follow-up 1 year after delivery
  Systolic and diastolic blood pressure will be measured with the participant in sitting position and with average of three readings measured with two minute intervals.
Change in total cholesterol and LDL | Measured at baseline and at follow-up 1 year after delivery
  Blood samples will be drawn after an overnight fast and will include measures of lipids
Impaired fasting glucose (IFG) and impaired glucose tolerance (IGT) | Measured at baseline and at follow-up 1 year after delivery
  IFG and IGT will be assessed based on the glucose measurements
Change in physical health quality of life | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire. Quality of life will be measured using the 12-item Short Form Health Survey (SF-12v2). Summary score will be calculated for the physical health domain. The SF-12 summary score ranges from 0 to 100, with higher scores representing better self-reported quality of life/health.
Change in walking patterns physical activity | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire. Physical activity will be measured using adapted version of the International Physical Activity Questionnaire (IPAQ) short form. Physical activity levels will be measured in minutes per week.
Differences in breastfeeding duration | Measured at follow-up 1 year after delivery
  Assessed through questionnaire.
Changes in social support for diet and exercise | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire.Will be measured using the Social Support and Eating Habits and Social Support and Exercise scales. Higher scores indicate more social support.
Changes in exercise self-regulation and motivation | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire.Will be measured using the TSRQ. Higher scores indicate higher self-regulation and motivation.
Change in self-efficacy | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire.Will be measured using the General Self-efficay scale. Higher scores indicate higher self-efficay.
Changes in risk perception | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire.Will be measured using the RPS-DD questionnaire.
Changes in health literacy | Measured at baseline and at follow-up 1 year after delivery
  Assessed through questionnaire.Will be measured using the HLQ. Higher scores indicate higher health literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Terkildsen Maindal, MPH, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim C, Newton KM, Knopp RH. Gestational diabetes and the incidence of type 2 diabetes: a systematic review. Diabetes Care. 2002 Oct;25(10):1862-8. doi: 10.2337/diacare.25.10.1862. PMID 12351492
- [Background] Ratner RE, Christophi CA, Metzger BE, Dabelea D, Bennett PH, Pi-Sunyer X, Fowler S, Kahn SE; Diabetes Prevention Program Research Group. Prevention of diabetes in women with a history of gestational diabetes: effects of metformin and lifestyle interventions. J Clin Endocrinol Metab. 2008 Dec;93(12):4774-9. doi: 10.1210/jc.2008-0772. Epub 2008 Sep 30. PMID 18826999
- [Background] Stage E, Ronneby H, Damm P. Lifestyle change after gestational diabetes. Diabetes Res Clin Pract. 2004 Jan;63(1):67-72. doi: 10.1016/j.diabres.2003.08.009. PMID 14693414
- [Derived] Jensen NH, Kragelund Nielsen K, Dahl-Petersen IK, Kampmann U, Damm P, Ovesen P, Mathiesen ER, Vinter CA, Davidsen E, Thogersen M, Timm A, Andersen LLT, Knorr S, Jensen DM, Maindal HT. Health promotion intervention among women with recent gestational diabetes mellitus: penetration, participation, and baseline findings from the Face-it randomized controlled trial. BMJ Open Diabetes Res Care. 2023 Oct;11(5):e003529. doi: 10.1136/bmjdrc-2023-003529. PMID 37793679
- [Derived] Maindal HT, Timm A, Dahl-Petersen IK, Davidsen E, Hillersdal L, Jensen NH, Thogersen M, Jensen DM, Ovesen P, Damm P, Kampmann U, Vinter CA, Mathiesen ER, Nielsen KK. Systematically developing a family-based health promotion intervention for women with prior gestational diabetes based on evidence, theory and co-production: the Face-it study. BMC Public Health. 2021 Sep 3;21(1):1616. doi: 10.1186/s12889-021-11655-2. PMID 34479526
- [Derived] Nielsen KK, Dahl-Petersen IK, Jensen DM, Ovesen P, Damm P, Jensen NH, Thogersen M, Timm A, Hillersdal L, Kampmann U, Vinter CA, Mathiesen ER, Maindal HT; Face-it Study Group. Protocol for a randomised controlled trial of a co-produced, complex, health promotion intervention for women with prior gestational diabetes and their families: the Face-it study. Trials. 2020 Feb 7;21(1):146. doi: 10.1186/s13063-020-4062-4. PMID 32033613

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT03997773/SAP_000.pdf